CLINICAL TRIAL: NCT03628586
Title: Can a Multi-marker Strategy Improve Risk Stratification and Expedite Discharge in Unstable Angina? A Comparison With High Sensitive Troponin T
Brief Title: Biomarkers and Risk Scores for Risk Stratification of Unstable Angina
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Liverpool University Hospitals NHS Foundation Trust (Other Government)
Collaborators: University of Liverpool (Other)
Responsible Party: Principal Investigator, Aleem Khand, consultant interventional cardiologist, Liverpool University Hospitals NHS Foundation Trust
Other Study IDs: AintreeNHS1
Record Dates: First submitted 2018-08-09; First posted 2018-08-14 (Actual); Last update posted 2018-08-17 (Actual); Status verified 2018-08

CONDITIONS: Chest Pain
Keywords: acute coronary syndrome; biomarkers, HS troponins
MeSH Terms: conditions — Chest Pain; Acute Coronary Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — plasma samples to allow extraction for a range of biologically plausible biomarkers associated with elevated risk in suspected acute coronary syndromes
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The main purpose of the study is to improve management and expedite safe discharge of patients presenting with chest pain with troponin ≤14ng/l using fifth generation, 'highly sensitive' troponin T. Our aim would be to specifically test in a prospective study whether biomarkers for left ventricular wall stress (NT pro brain natriuretic peptide), ischaemia (Heart-type fatty acid protein) and a novel marker of stress, raised in a number of pathological states growth differentiation factor -15, add significantly to the prognostic value of clinical information and resting ECG presenting with ischaemic sounding chest pain. The 5th generation troponin assay will be used and the range of values from 1-14ng/l will also be compared to the biomarkers studied in terms of hard cardiac endpoints. Recent studies have indicated that very low levels of detected troponin in patients with stable coronary artery disease do adversely impact on cardiac death and the development of heart failure.

DETAILED DESCRIPTION:
Chest pain accounts for up to 1% of visits to GPs in England, about 700000 visits (5%) to emergency departments and up to 25% of emergency admissions to hospitals. Recent epidemiological studies indicate a substantial and increasing rate of admissions with chest pain even as admissions with acute myocardial infarction are falling. From 1986 to 2000 the rate of admissions for chest pain in Scottish hospitals more than doubled. Further work by the same group indicates that admission to hospital with angina, excluding those coded for acute coronary syndrome or acute myocardial infarction, is associated with a 30 day mortality of 1.5%. Other studies have identified a sizable event rate in patients who have been 'troponin negative'. This increasing phenomenon places great strain on the NHS and indeed any health provider. Any form of testing that adds significant incremental value to established tests and that can effectively rule out myocardial ischaemia and moreover demonstrate good medium and long-term outcome could potentially benefit both patients and the NHS delivery of healthcare.

Brain Natriuretic Peptide Biochemical markers of left ventricular wall stress or ischaemia could enhance the diagnostic accuracy of exercise tolerance tests. These have been used successfully for the detection of left ventricular dysfunction, heart failure and in the risk stratification of acute coronary syndromes.

Biomarkers of acute stress

Growth Differentiation Factor -15 Transforming growth Factor constitute a superfamily of cytokines that exert prominent actions in adult haemostasis and adaptation by regulating cell survival, proliferation and differentiation. GDF-15 is a distant member of the TGF-B superfamily. In animal models it is induced in response to ischaemia-reperfusion injury, pressure overload and heart failure possibly via pro-inflammatory cytokine and oxidative stress dependent signalling pathways. There is both evidence of an adverse outcome in patients with an elevated GDF-15 level in highly selected trials with NSTEMI as well as the non-selected chest pain population. This latter analysis was a post-hoc one and there are no prospective studies in an unselected chest pain population evaluating GDF-15.

Heart Type Fatty Acid Binding Protein (HFABP)- Direct evidence of myocardial ischaemia HFAP is a low molecular weight protein that is involved in the intracellular uptake and buffering of free fatty acids in the myocardium. It has been shown to be a sensitive and early marker of myocardial infarction providing direct evidence of myocardial ischaemia as well as myocyte necrosis unlike HSCRP and BNP. This is intuitive given its small molecular size and consequently its propensity to be leaked from the porous membranes of ischaemic myocardial cells. In the study by Kilcullen et al even Tn negative patients were well stratified by HFABP.

The role of inflammation and specifically HS-CRP Inflammatory processes play an integral part in the process of atherogenesis and atherothrombosis. There is clear evidence of their involvement in the processes that lead to the development of intermediate and mature atheromatous plaques. Inflammatory cells and mediators are also clearly implicated in the final breach between the thin fibrous cap and circulating platelets and coagulation proteins. Several mediators have been investigated. These include HS-CRP, serum amyloid A, myeloperoxidase and interleukin-6. They are detectable in a large proportion of patients with ACS including those with no evidence of myocyte necrosis. It is not clear if these markers directly contribute to the pathology of plaque destabilisation and ischaemia or whether they are largely a 'byproduct' of the inflammation engendered by ischaemia and plaque rupture. CRP promotes uptake of LDL cholesterol by monocytes, induces the production of tissue factor, activates complement within arterial plaque as well as stimulating the expression of adhesion molecules. In this regard at least it maybe postulated that CRP is a direct participant in atherothrombosis. It has also been demonstrated that the measurement of Hs-CRP can grant additional prognostic information to patients with negative serial cardiac troponins. However both of these studies were post-hoc sub-studies of randomised controlled trials. Posthoc analyses of the PROSPER study however indicated that measurement oinf HS-CRP added only a small incremental prognostic value to patients at risk of vascular events. Recent results of the Jupiter study gives rise for hope that inflammation as determined by CRP can improve outcome if used a therapeutic decision tool for rosuvastatin treatment in patients who do not fulfil criteria for primary treatment of hyperlipidaemia. This does suggest the potential value of therapeutic decision making with HS-CRP albeit in a different setting.

Rationale for study In consecutive series of patients admitted with troponin negative chest pain the investigators aim to evaluate the independent prognostic value of resting NT-pro BNP, basal HFABP, GDF-15 and HS-CRP. The relationship of these markers to long term hard endpoints will be investigated . The investigators aim to specifically assess whether alone or in combination these can aid in the risk stratification of acute chest pain admissions that do not have evidence for myocyte necrosis. A range of parameters such as the presence of anaemia, ECG changes and pain characteristics will be included in a model to assess the tested parameters relative effect and relationship with clinical outcome. The aim is to define the independent, cumulative incremental benefit of resting NT-pro BNP, resting HFABP, GDF-15 and HS-CRP and to determine whether either alone or in combination this information may help improve risk stratification and ultimately therapeutic decision making in patients with troponin negative chest pain.

ELIGIBILITY:
Inclusion Criteria:

* Patients presenting within 12 hours of chest pain thought to be cardiac in origin but with no ST segment elevation on ECG
* 5th generation troponin T <15ng/l
* Consent for inclusion in study and consent for follow-up over 3 years either by telephone or GP contact

Exclusion Criteria:

* Troponin positive patients, Tn T>=15ng/lµg/l
* Diagnosis of non-cardiac chest pain made at outset
* Known History of chronic heart failure or cardiomyopathy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 1. Admission with chest pain which could be due to underlying ischaemic heart disease
  2. HSTroponin T < 15ng/L in patients with possible ischaemic sounding chest pain admitted to hospital at least 6 hours since onset of chest pain or in those with pain <3hours since admission with no STEMI, a baseline HStroponin T <15ng/l (time 0 on admission) and HSTroponin T <15ng/l at 3 hours and <20% increase compared to baseline (time 0)
  3. Ability to give informed consent for extraction of blood for biochemical screening
Sampling Method: Non-Probability Sample
Enrollment: 489 (Actual)
Dates: Start 2011-01-10 (Actual); Primary Completion 2018-10-01 (Estimated); Study Completion 2018-12-01 (Estimated)

PRIMARY OUTCOMES:
Major Adverse Cardiac Event: death, myocardial infarction, revascularisation | 3 years
  All cause death, myocardial infarction and revascularisation within 3 years of index presentation

IPD SHARING:
Plan to Share IPD: Undecided
we currently are focused on completing extensive follow-up and hope to make database available to reviewers and journal editors

REFERENCES:
- [Derived] Jones J, Hughes E, Dobson R, Ashrafi R, Heseltine T, Campbell M, Collinson P, Khand A. Risk Stratification of Acute Chest Pain in Patients With High-Sensitivity Troponin T Below the 99th Percentile: A Long-Term Cohort Study Assessing the Incremental Value of Necrosis and Non-necrosis Biomarkers to Clinical Risk Scores. J Am Heart Assoc. 2025 Oct 21;14(20):e040590. doi: 10.1161/JAHA.124.040590. Epub 2025 Oct 14. PMID 41085181